CLINICAL TRIAL: NCT02772107
Title: Temozolomide as Maintenance Therapy Following Induction Chemotherapy in Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, yihu, chief of oncology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301PLAGH
Record Dates: First submitted 2016-05-07; First posted 2016-05-13 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BSC group (Experimental): Patients in the study will receive the following for the duration of the study:First-line chemotherapy according to the NCCN guidelines. The study will consist of 21-day cycles, to a maximum of 6 cycles of therapy for the first-line chemotherapy. Radiotherapy was allowed. Follow-up until disease progression.
  Interventions: Drug: first-line chemotherapy; Radiation: Prophylactic cranial irradiation; Radiation: thoracic radiotherapy
- TMZ group (Experimental): Patients will receive platinum-based first-line chemotherapy according to the NCCN guidelines. The study will consist of 21-day cycles, to a maximum of 6 cyclesfor the first-line chemotherapy. After first-line treatment, temozolomide will be given alone as maintenance therapy in all patients who have achieved study entry hematologic criteria and who do not have progressive disease or severe toxicity. During temozolomide maintenance therapy, patients will receive temozolomide at 150mg/m2/d for 5 days of a 28-day cycle orally daily. Temozolomide maintenance therapy will continue until progressive disease or irreversible toxicity occurs.
  Re-staging will be performed every 2 cycles (every 8 weeks) during the study, radiotherapy was allowed.
  Interventions: Drug: Temozolomide; Drug: first-line chemotherapy; Radiation: Prophylactic cranial irradiation; Radiation: thoracic radiotherapy

INTERVENTIONS:
Drug: Temozolomide — Temozolomide is a nonclassic oral alkylating agent. Temozolomide will be given alone as maintenance therapy in patients who have achieved study entry hematologic criteria and who do not have progressive disease or severe toxicity. During temozolomide maintenance therapy, patients will receive temozolomide at 150mg/m2/d for 5 days of a 28-day cycle orally daily. Temozolomide maintenance therapy will continue until progressive disease or irreversible toxicity occurs.
  Arms: TMZ group
Drug: first-line chemotherapy — first-line chemotherapy must be platinum-based: cisplatin(75mg/m2 for d1) or carboplatin（AUC 5 for d1) combined with etoposide（100mg/m2 for d1-d3）
Radiation: Prophylactic cranial irradiation — Prophylactic cranial irradiation was allowed if necessary
Radiation: thoracic radiotherapy — thoracic radiotherapy was allowed if necessary

SUMMARY:
Temozolomide may delay progression in sequence with chemotherapy. This open-label, randomized,multicenter phase II trial was designed to evaluate the role of Temozolomide following 4 or 6 cycles of platinum-based first-line chemotherapy in patients with newly diagnosed estensive-stage SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically and/or histologically confirmed small-cell lung cancer with extensive-stage disease
* Patients must have measurable disease, this can include brain metastases
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate bone marrow function, as defined by: absolute neutrophil count (ANC) >1,500/µL; platelets >100,000/µL; hemoglobin >=9.0 g/dL
* Normal organ function, defined as follows: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5 × the upper limit of normal (ULN), or AST and ALT <=5 × the ULN if liver function abnormalities are due to underlying malignancy; total serum bilirubin <=1.5 × the ULN; serum creatinine <=1.5 × the ULN
* the time interval from the data of the last chemotherapy to random must be between 3 and 7 weeks
* Women of childbearing potential and men with partners of childbearing potential must agree to use a form of birth control that is acceptable to their physician to prevent pregnancy during treatment
* Patients must be informed of the investigational nature of this study and sign an informed consent form

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients receiving other investigational agents
* Patients with leptomeningeal involvement
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition or HIV-positive patients on combination antiretroviral therapy. However, HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because these patients are at increased risk of lethal infections when treated with marrow- suppressive therapy. Excluding patients on HAART is necessary due to the potential for pharmacokinetic interactions with temozolomide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
PFS of the maintenance therapy | 2 years
  from the data of randomized to the date of disease progression or the patient dies

SECONDARY OUTCOMES:
PFS | 2 years
  from the date of first-line chemotherapy to the date of disease progression
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided